CLINICAL TRIAL: NCT02690103
Title: Clinical Study of a Biological Response Modifier (Arabinoxylan Rice Bran/MGN-3/Biobran) With Interferon-Alpha for the Treatment of Hepatitis C Infection
Brief Title: Response Modifier (Arabinoxylan Rice Bran/MGN-3/Biobran) With Interferon-Alpha for HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Daiwa Pharmaceutical Corporation Co, Ltd, Tokyo 154-0024 Japan (Unknown); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hosny Salama, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2016-02-08; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Arabinoxylan; HCV; Viremia; Biobran; PEG interferon
MeSH Terms: conditions — Hepatitis C, Chronic; Viremia | interventions — polysaccharide MGN3; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Patients are treated with 180µg of pegylated IFN (Pegasys-Roche) subcutaneously weekly for three months. In addition, they are given ribavirin according to their body weight (1200 mg for those over 75 kg and 1000 mg for those under 75 kg).
  Interventions: Drug: pegylated IFN; Drug: Ribavirin
- Group 2 (Experimental): Patients are treated with Biobran, at a dose of 1g per day, allocated in packets, taken orally with meals for the three months duration of the study. Biobran is a denatured hemicellulose that is obtained by reacting rice bran hemicellulose with multiple carbohydrate hydrolyzing enzymes from Shiitake mushrooms. It is a polysaccharide that contains ß-1, 3-glucans, and activated hemicellulose.
  Interventions: Dietary Supplement: Biobran

INTERVENTIONS:
Drug: pegylated IFN — Patients are treated with 180µg of pegylated IFN (Pegasys-Roche) subcutaneously weekly for three months.
  Arms: Group 1
Dietary Supplement: Biobran — Biobran, at a dose of 1g per day, allocated in packets, taken orally with meals for the three months duration of the study. Biobran is a denatured hemicellulose that is obtained by reacting rice bran hemicellulose with multiple carbohydrate hydrolyzing enzymes from Shiitake mushrooms. It is a polysaccharide that contains ß-1, 3-glucans, and activated hemicellulose. Biobran was kindly provided by Daiwa Pharmaceuticals Co. Ltd., Tokyo, Japan.
  Arms: Group 2
Drug: Ribavirin — Ribavirin is prescribed according to patients body weight (1200 mg for those over 75 kg and 1000 mg for those under 75 kg).
  Arms: Group 1

SUMMARY:
Current treatments for Hepatitis C virus (HCV) have severe side effects and are very expensive. There is a need to explore effective natural therapies against HCV that are less toxic and more cost-effective.

37 chronic HCV infected patients were randomized into two groups and treated with PEG interferon plus ribavirin for the first group or Biobran, an arabinoxylan from rice bran (1 g/day) for the second group. Viremia level, liver enzymes, γ-interferon (IFN-γ) levels in serum, and toxicity were checked before and three months after treatment.

DETAILED DESCRIPTION:
The current study is a preliminary investigation of whether Biobran has the ability to restrict viremia in patients with chronic HCV or not. In addition, we examined the effect of Biobran on liver enzymes and inflammation as well as assessing any side effects of Biobran. Results show that treatment with Biobran resulted in a significant reduction in the viral load, an increase in liver enzymes, and patients reported good health.

For the randomized trial, we selected 37 patients who had been admitted to El-Kasr El-Aini Hospital at Cairo, Egypt. The patients had been diagnosed with genotype 4 HCV infection. The study was approved by Cairo University Hospital, Cairo, Egypt and by IRB at Charles Drew school of medicine and Science, Los Angeles, CA, USA. The study protocol conformed to the ethical guidelines of the 1975 Declaration of Helsinki as reflected in the prior approval by Cairo University, El-Kasr El-Aini Hospital, Cairo, Egypt and by the Institutional Review Board (IRB) at Cairo University, Egypt and Charles R Drew University (CDU), Los Angeles, CA., USA.

Thirty-seven patients of both sexes (23 males and 14 females) with HCV (genotype 4), between the ages of 15 and 69, participated in the current study. Informed consent was obtained from all participants.

The patients were divided randomly into two groups: the Biobran group and the PEG interferon plus ribavirin (control) group . Prior to treatment, clinical characteristics were determined for the patients in each group. The clinical characteristics of the HCV patients were investigated for hepatitis C, alpha-fetoprotein (AFP) levels, total leucocyte count (TLC), Platelet (PLT) count, Hemoglobin (Hb) levels, triglyceride (TG) levels, glycated hemoglobin (HbA1c) levels, blood clotting using International Normalized Ratio (INR), creatinine per milliliter (Cr/ml), and random blood sugar (RBG).

Patients in the control group were treated with 180µg of pegylated IFN (Pegasys-Roche) subcutaneously weekly for three months. In addition, they were given ribavirin according to their body weight (1200 mg for those over 75 kg and 1000 mg for those under 75 kg). The Biobran group was treated with Biobran, at a dose of 1g per day, allocated in packets, taken orally with meals for the three months duration of the study. Biobran is a denatured hemicellulose that is obtained by reacting rice bran hemicellulose with multiple carbohydrate hydrolyzing enzymes from Shiitake mushrooms. It is a polysaccharide that contains ß-1, 3-glucans, and activated hemicellulose. Biobran was kindly provided by Daiwa Pharmaceuticals Co. Ltd., Tokyo, Japan.

The patients were divided randomly into two groups: the Biobran group and the PEG interferon plus ribavirin (control) group . Prior to treatment, clinical characteristics were determined for the patients in each group. The clinical characteristics of the HCV patients were investigated for hepatitis C, alpha-fetoprotein (AFP) levels, total leucocyte count (TLC), Platelet (PLT) count, Hemoglobin (Hb) levels, triglyceride (TG) levels, glycated hemoglobin (HbA1c) levels, blood clotting using International Normalized Ratio (INR), creatinine per milliliter (Cr/ml), and random blood sugar (RBG).

Viral load levels, toxicity, liver enzymes, and γ-interferon (IFN-γ) levels were examined before and three months after treatment. Viral load was examined by quantitative polymerase chain reaction (PCR) test using COBAS® TaqMan® Analyzer (Roche Corporation). IFN-γ, AFP, ALT, and AST levels were analyzed using specific Elisa Kits, which were performed by Spectrum Chemical Manufacturing Corporation, Gardena, CA, USA, and toxicity was assessed by a questionnaire, physician observation, and laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic HCV infection and chronic active liver diseases.

Exclusion Criteria:

* Patients diagnosed with chronic HBV , HIV infection , autoimmune disorders , any heart diseases , any kidney diseases or any blood disease , any neoplastic disorders.
* Pregnant or lactating ladies , and drug abusers will be excluded.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of BioBran on the viraemia levels in chronic HCV infected patients | 3-month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hosny Salama, MD, Principal Investigator — Cairo University, Egypt; Abdel Rahaman Zekry, PhD, Study Director — Cairo University, Egypt; Mamdouh Ghoneum, MD, Principal Investigator — University of California , Los Angeles, USA; Tarneem Darwish, MD, Study Chair — Cairo University , Egypt; Dalia Omran, MD, Study Chair — Cairo University , Egypt; Rasha Ahmed, MD, Study Chair — Cairo University , Egypt; Sherif Mousa, MD, Study Chair — Cairo University , Egypt; Sherine Abdel alim, MD, Study Chair — Cairo University , Egypt; Hany Khattab, MD, Study Chair — Cairo University , Egypt; Mervat Al Ansary, MD, Study Chair — Cairo University , Egypt; Nemat Kasem, MD, Study Chair — Cairo University , Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] University of Washington/Seattle STD/HIV Prevention Training Center. Hepatitis Web Study. 2013. Available at: http://www.cdc.gov/hepatitis/Resources/Professionals/PDFs/ABCTable.pdf. Accessed 29 November 2015.
- [Background] Sievert W, Altraif I, Razavi HA, Abdo A, Ahmed EA, Alomair A, Amarapurkar D, Chen CH, Dou X, El Khayat H, Elshazly M, Esmat G, Guan R, Han KH, Koike K, Largen A, McCaughan G, Mogawer S, Monis A, Nawaz A, Piratvisuth T, Sanai FM, Sharara AI, Sibbel S, Sood A, Suh DJ, Wallace C, Young K, Negro F. A systematic review of hepatitis C virus epidemiology in Asia, Australia and Egypt. Liver Int. 2011 Jul;31 Suppl 2:61-80. doi: 10.1111/j.1478-3231.2011.02540.x. PMID 21651703
- [Background] Lavanchy D. Evolving epidemiology of hepatitis C virus. Clin Microbiol Infect. 2011 Feb;17(2):107-15. doi: 10.1111/j.1469-0691.2010.03432.x. PMID 21091831
- [Background] Ghoneum M. Anti-HIV activity in vitro of MGN-3, an activated arabinoxylane from rice bran. Biochem Biophys Res Commun. 1998 Feb 4;243(1):25-9. doi: 10.1006/bbrc.1997.8047. PMID 9473473
- [Background] Ghoneum M. Enhancement of human natural killer cell activity by modified arabinoxylane from rice bran (MGN-3). Int J Immunotherapy 1998; XIV(2):89-99.
- [Background] Ghoneum M, Abedi S. Enhancement of natural killer cell activity of aged mice by modified arabinoxylan rice bran (MGN-3/Biobran). J Pharm Pharmacol. 2004 Dec;56(12):1581-8. doi: 10.1211/0022357044922. PMID 15563765
- [Background] Cholujova D, Jakubikova J, Czako B, Martisova M, Hunakova L, Duraj J, Mistrik M, Sedlak J. MGN-3 arabinoxylan rice bran modulates innate immunity in multiple myeloma patients. Cancer Immunol Immunother. 2013 Mar;62(3):437-45. doi: 10.1007/s00262-012-1344-z. Epub 2012 Sep 2. PMID 22941038
- [Background] Perez-Martinez A, Valentin J, Fernandez L, Hernandez-Jimenez E, Lopez-Collazo E, Zerbes P, Schworer E, Nunez F, Martin IG, Sallis H, Diaz MA, Handgretinger R, Pfeiffer MM. Arabinoxylan rice bran (MGN-3/Biobran) enhances natural killer cell-mediated cytotoxicity against neuroblastoma in vitro and in vivo. Cytotherapy. 2015 May;17(5):601-12. doi: 10.1016/j.jcyt.2014.11.001. Epub 2014 Dec 23. PMID 25541298
- [Background] Cholujova D, Jakubikova J, Sedlak J. BioBran-augmented maturation of human monocyte-derived dendritic cells. Neoplasma. 2009;56(2):89-95. doi: 10.4149/neo_2009_02_89. PMID 19239320
- [Background] Ghoneum M, Agrawal S. Activation of human monocyte-derived dendritic cells in vitro by the biological response modifier arabinoxylan rice bran (MGN-3/Biobran). Int J Immunopathol Pharmacol. 2011 Oct-Dec;24(4):941-8. doi: 10.1177/039463201102400412. PMID 22230400
- [Background] Ghoneum M, Agrawal S. Mgn-3/biobran enhances generation of cytotoxic CD8+ T cells via upregulation of dec-205 expression on dendritic cells. Int J Immunopathol Pharmacol. 2014 Oct-Dec;27(4):523-30. doi: 10.1177/039463201402700408. PMID 25572732
- [Background] Ghoneum M, Jewett A. Production of tumor necrosis factor-alpha and interferon-gamma from human peripheral blood lymphocytes by MGN-3, a modified arabinoxylan from rice bran, and its synergy with interleukin-2 in vitro. Cancer Detect Prev. 2000;24(4):314-24. PMID 11059563
- [Background] Noaman E, Badr El-Din NK, Bibars MA, Abou Mossallam AA, Ghoneum M. Antioxidant potential by arabinoxylan rice bran, MGN-3/biobran, represents a mechanism for its oncostatic effect against murine solid Ehrlich carcinoma. Cancer Lett. 2008 Sep 18;268(2):348-59. doi: 10.1016/j.canlet.2008.04.012. Epub 2008 Jun 12. PMID 18554778
- [Background] Ghoneum M, Badr El-Din NK, Abdel Fattah SM, Tolentino L. Arabinoxylan rice bran (MGN-3/Biobran) provides protection against whole-body gamma-irradiation in mice via restoration of hematopoietic tissues. J Radiat Res. 2013 May;54(3):419-29. doi: 10.1093/jrr/rrs119. Epub 2013 Jan 3. PMID 23287771
- [Background] Ghoneum M. Anti-HIV activity by MGN-3 in vitro. XI International Conference on AIDS. Vancouver, July 7-12, 1996.
- [Background] Tazawa K, Ichihashi K, Fuji T, Omura K, Anazawa M, Maeda H. The orally administration of the Hydrolysis Rice Bran prevents a common cold syndrome for the elderly people based on the immunomodulatory function. J Trad Med 2003; 20:132-41.
- [Background] Caroleo B, Gallelli L, Staltari O, De Sarro G, Guadagnino V. Serum transaminase elevations during pegylated interferon treatment of chronic HCV hepatitis probably induced by polyethylene glycol. Intervirology. 2008;51(6):407-9. doi: 10.1159/000205266. Epub 2009 Mar 4. PMID 19258719
- [Background] Kleppinger EL, Ragan AP. Elevated hepatic transaminases associated with the use of interferon alfacon-1 and ribavirin. Am J Health Syst Pharm. 2009 Mar 1;66(5):465-8. doi: 10.2146/ajhp080243. PMID 19233994
- [Background] Levent G, Ali A, Ahmet A, Polat EC, Aytac C, Ayse E, Ahmet S. Oxidative stress and antioxidant defense in patients with chronic hepatitis C patients before and after pegylated interferon alfa-2b plus ribavirin therapy. J Transl Med. 2006 Jun 20;4:25. doi: 10.1186/1479-5876-4-25. PMID 16787540
- [Background] Tatsumi T, Takehara T, Miyagi T, Nakazuru S, Mita E, Kanto T, Hiramatsu N, Hayashi N. Hepatitis C virus-specific CD8+ T cell frequencies are associated with the responses of pegylated interferon-alpha and ribavirin combination therapy in patients with chronic hepatitis C virus infection. Hepatol Res. 2011 Jan;41(1):30-8. doi: 10.1111/j.1872-034X.2010.00734.x. Epub 2010 Oct 7. PMID 21040277
- [Background] Sreenarasimhaiah J, Jaramillo A, Crippin J, Lisker-Melman M, Chapman WC, Mohanakumar T. Concomitant augmentation of type 1 CD4+ and CD8+ T-cell responses during successful interferon-alpha and ribavirin treatment for chronic hepatitis C virus infection. Hum Immunol. 2003 May;64(5):497-504. doi: 10.1016/s0198-8859(03)00041-7. PMID 12691700
- [Background] Baranova I, Vishnyakova T, Bocharov A, Chen Z, Remaley AT, Stonik J, Eggerman TL, Patterson AP. Lipopolysaccharide down regulates both scavenger receptor B1 and ATP binding cassette transporter A1 in RAW cells. Infect Immun. 2002 Jun;70(6):2995-3003. doi: 10.1128/IAI.70.6.2995-3003.2002. PMID 12010990
- [Background] Rice CM. New insights into HCV replication: potential antiviral targets. Top Antivir Med. 2011 Aug-Sep;19(3):117-20. PMID 21946389
- [Background] Alter HJ, Liang TJ. Hepatitis C: the end of the beginning and possibly the beginning of the end. Ann Intern Med. 2012 Feb 21;156(4):317-8. doi: 10.7326/0003-4819-156-4-201202210-00014. No abstract available. PMID 22351718
- [Background] Park Y, Pham TX, Lee J. Lipopolysaccharide represses the expression of ATP-binding cassette transporter G1 and scavenger receptor class B, type I in murine macrophages. Inflamm Res. 2012 May;61(5):465-72. doi: 10.1007/s00011-011-0433-3. Epub 2012 Jan 13. PMID 22240665
- [Background] Scheel TK, Rice CM. Understanding the hepatitis C virus life cycle paves the way for highly effective therapies. Nat Med. 2013 Jul;19(7):837-49. doi: 10.1038/nm.3248. PMID 23836234
- [Background] Frese M, Schwarzle V, Barth K, Krieger N, Lohmann V, Mihm S, Haller O, Bartenschlager R. Interferon-gamma inhibits replication of subgenomic and genomic hepatitis C virus RNAs. Hepatology. 2002 Mar;35(3):694-703. doi: 10.1053/jhep.2002.31770. PMID 11870386
- [Background] Schmidt J, Blum HE, Thimme R. T-cell responses in hepatitis B and C virus infection: similarities and differences. Emerg Microbes Infect. 2013 Mar;2(3):e15. doi: 10.1038/emi.2013.14. Epub 2013 Mar 27. PMID 26038456
- [Derived] Salama H, Medhat E, Shaheen M, Zekri AN, Darwish T, Ghoneum M. Arabinoxylan rice bran (Biobran) suppresses the viremia level in patients with chronic HCV infection: A randomized trial. Int J Immunopathol Pharmacol. 2016 Dec;29(4):647-653. doi: 10.1177/0394632016674954. Epub 2016 Oct 31. PMID 27799299